CLINICAL TRIAL: NCT05125627
Title: Randomized, Two-sequence, Two-treatment, Four-period, Open Label, Single Dose, Crossover, Intravaginal Bioequivalence Study of 200 mg Soft Capsule Progesterone vs Utrogestan® in Healthy Female Subjects Under Fasting Conditions.
Brief Title: Fasting Bioequivalence Study of 2 Progesterone Soft Capsules 200 mg in 66 Healthy Female Subjects Under Vaginal Route
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Joint Stock Company "Farmak" (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: FK/BE/PGIV/19
Record Dates: First submitted 2021-11-08; First posted 2021-11-18 (Actual); Last update posted 2021-11-18 (Actual); Status verified 2021-11

CONDITIONS: Pharmacokinetics
Keywords: bioequivalence; pharmacokinetics; generic drugs; Progesterone; Soft Capsule
MeSH Terms: interventions — Progesterone; Utrogestan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment A (Experimental): Progesterone 200 mg Soft Capsule (JSC "Farmak", Ukraine)
  Each dose was administered Intravaginally, the capsule introduced deeply into the vagina while lying down, after at least 10 hrs of fasting, under the direct supervision of the Principal and/ or clinical Investigator
  Interventions: Drug: Progesterone 200 mg Soft Capsule (JSC "Farmak", Ukraine)
- Treatment B (Active Comparator): Utrogestan® 200 mg Soft Capsule (Manufacturer: Cyndea Pharma, S.L., Spain, MAH: Laboratoires Besins International, France)
  Each dose was administered Intravaginally, the capsule introduced deeply into the vagina while lying down, after at least 10 hrs of fasting, under the direct supervision of the Principal and/ or clinical Investigator
  Interventions: Drug: Utrogestan® 200 mg Soft Capsule (Manufacturer: Cyndea Pharma, S.L., Spain, MAH: Laboratoires Besins International, France)

INTERVENTIONS:
Drug: Progesterone 200 mg Soft Capsule (JSC "Farmak", Ukraine) — Each dose was administered Intravaginally, the capsule introduced deeply into the vagina while lying down, after at least 10 hrs of fasting, under the direct supervision of the Principal and/ or clinical Investigator
  Other Names: Injesta
  Arms: Treatment A
Drug: Utrogestan® 200 mg Soft Capsule (Manufacturer: Cyndea Pharma, S.L., Spain, MAH: Laboratoires Besins International, France) — Each dose was administered Intravaginally, the capsule introduced deeply into the vagina while lying down, after at least 10 hrs of fasting, under the direct supervision of the Principal and/ or clinical Investigator
  Other Names: Utrogestan®
  Arms: Treatment B

SUMMARY:
This study was designed to assess the bioequivalence of Progesterone 200 mg Soft Capsule (JSC "Farmak", Ukraine) versus Utrogestan® 200 mg Soft Capsule (Manufacturer: Cyndea Pharma, S.L., Spain, MAH: Laboratoires Besins International, France) after a single Vaginal dose in healthy female subjects under fasting conditions.

DETAILED DESCRIPTION:
An open-label, randomized, single dose, two-treatment, four-period, two-sequence, fully replicated crossover bioequivalence study with a washout period of 7 days in healthy female subjects under fasting conditions.Mode of administration:Intravaginally, the capsule introduced deeply into the vagina while lying down.During each period 25 blood samples were drawn 5 mL at (-1.00,-0.50,-0.137), before dosing and at 0.50, 1.00, 1.50, 2.00,2.50, 3.00, 3.50, 4.00, 4.50, 5.00, 5.50, 6.00, 7.00, 8.00, 9.00, 10.00, 12.00, 16.00, 24.00,36.00, 48.00, and 72.00 hours after dosing.

ELIGIBILITY:
Inclusion Criteria:

* Non-smoker or past-smoker (an ex-smoker is defined as someone who has completely stopped using nicotine products, including nicotine cessation therapy, for at least 180 days prior to the first study drug administration).
* Body Mass Index (BMI) ≥18.5 and ≤ 30 kg/m2, inclusive and body weight between 45 kg and 100 kg(on the day of screening).
* Subject is available for the whole study and has provided her written informed consent
* Subjects in good health, as determined by screening medical history, physical examination, vital signs assessments (pulse rate, systolic and diastolic blood pressure, and body temperature) and 12-lead electrocardiogram (ECG) . Minor deviations outside the reference ranges will be acceptable, if deemed not clinically significant by the Investigator.
* Acceptance of use of contraceptive measures during the whole study.
* Normal Liver and kidney function tests (on Screening)
* All laboratory screening results within the normal range, or deemed clinically insignificant by Investigator.
* The thickness of the endothelial layer according to ultrasound of the pelvic organs is not less than 2 mm and not more than 4 mm (on Screening)

Exclusion Criteria:

* Known cardiovascular disease, history of hypotension
* History of gout, urolithiasis, nephrolithiasis and hyperuricaemia
* Gastrointestinal diseases, including gastric ulcer, renal or hepatic diseases and/or pathological findings present or in history, which might interfere with the drug pharmacokinetics.
* Known history or presence of food allergies, or any condition known to interfere with the absorption, distribution, metabolism or excretion of drugs.
* Acute or chronic diseases and/or clinical finding which may interfere with the aims of the study or with the drug's safety, tolerability, bioavailability and/or pharmacokinetics of the Investigational Medicinal Product (IMP).
* History of severe allergy or allergic reactions to the study IMP, its excipients or related drugs, wheat allergy history.
* Positive result of urine pregnancy test at screening or breast-feeding or lack of results of pregnancy test.
* Postponed acute diseases of the female genitals during the last 3 months, including vaginitis and / or vulvovaginitis.
* Chronic inflammatory and/or atrophic diseases of the pelvic organs.
* Benign neoplasms and anamnesis of hyperplastic processes, including mastopathy and endometrial hyperplasia.
* Surgical intervention on the pelvic organs, including hysterectomy, adnexectomy (It doesn't include the Subject who had a previous history of Cesarean section for 5 years or more provided that the Cesarean section was not for pathological reasons and/ or accompanied with cervix and uterus diseases or external genitals organs disease).
* Arterial or venous thromboembolism or thrombophlebitis in anamnesis.
* Reporting drug of abuse at screening
* Positive result of alcohol breath test at screening.
* The presence of nicotine or cotinine in urine at the screening.
* Serious mental disease and/or inability to cooperate with clinical team.
* Sitting blood pressure after a minimum of 5 minutes of rest is out of the range of 90-140 mmHg for systolic BP and/or 60-90 mmHg for diastolic BP and/or heart rate out of the range of 50-100 bpm during the screening procedure.
* Body temperature is out of the range of 35.7-37.6° C at screening.
* Orthostatic hypotension during the screening procedure or in the history.
* Reporting Drug, alcohol (of ≥ 40 g per day pure ethanol), solvents or caffeine abuse at screening.
* Getting a tattoo, body piercing or any cosmetic treatment involving skin piercing within 90 days before the screening unless evaluated by Investigator as non-significant for inclusion in the study.
* Donation of at least 400 ml of blood within 60 days, or more than 150 ml of blood within 30 days, or more than 100 ml blood plasma or platelets within 14 days before study Period I.
* Following a special diet (e.g. vegetarian) or dieting one month before the study initiation
* Allergy on peanut in anamnesis
* Less than 80 days between exit procedure in previous study and the first dosing in this study.
* Any significant clinical abnormality including Hepatitis B surface antigen (HBsAg), hepatitis C virus (HCV), and / or (human immunodeficiency virus) HIV. (On screening)
* Abnormal Kidney and/or Liver function tests and being assessed as clinically significant by the attending physician. (On screening).
* Results of laboratory tests are outside the normal range and being assessed as clinically significant by the attending physician (On screening).
* Previous liver disease or elevations in serum transaminases alanine aminotransferase (ALT) or aspartate aminotransferase AST ≥1.0 upper limit of normal (ULN) at the screening (ALT for women up to 63 U/L and AST up to 37 U/L).
* Any significant clinical abnormality, including a positive result of HBsAg and/or HCV and/or HIV test during screening procedure.
* Uric acid level for women > 6.0 mg/dl at the screening
* History of kidney disease with impaired renal function and level of creatinine in blood out of the normal laboratory range based on screening
* Anemia, hemoglobin below 12.0 g/L at screening.
* The intake of caffeine, xanthenes, or carbon dioxide (CO2)-containing beverages within 18 hours of drug administration
* Consumption of alcohol, grapefruit or grapefruit containing products within 7 days of drug administration.
* Ingestion of any supplements like vitamins or herbal products within 7 days prior to the initial dose of the study medication.
* Exhausting physical exercise in the last 48 hours (e.g. weight lifting) or any recent significant change in dietary or exercise habits.
* Abnormal Vital Signs and being assessed as clinically significant by the attending physician.
* Vomiting, Diarrhea on admission.
* Use of organ-toxic drugs or systemic drugs known to substantially alter liver metabolism within 90 days before the first dosing.
* Use of any prescription medication for a period of 14 days before the first dosing.
* Any systemic over-the-counter (OTC) drug treatment and/or vitamins and/or herbal treatment and/or food supplements within 14 days before the first dosing.
* Clinically significant illness within 28 days before the first dosing, including major surgery.
* Positive results of drug of abuse at check-in.
* Positive result of alcohol breath test at check-in.
* Reporting Drug, alcohol (of ≥ 40 g per day pure ethanol), solvents or caffeine abuse at check-in
* Positive urine pregnancy test at check-in.

Ages: 45 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — -Healthy postmenopausal females with amenorrhea duration of at least 6 months, but not more than 24 months.
Enrollment: 66 (Actual)
Dates: Start 2019-08-28 (Actual); Primary Completion 2019-10-21 (Actual); Study Completion 2019-10-21 (Actual)

PRIMARY OUTCOMES:
Cmax | up to 72 hours post-administration
  Cmax - Maximum plasma concentration derived/calculated from the concentrations of Progesterone Corrected determined in individual plasma samples for each subject
AUC0→last | up to 72 hours post-administration
  AUC0→last -The area under the plasma concentration-time curve

SECONDARY OUTCOMES:
Tmax | up to 72 hours post-administration
  Tmax -The time of the peak concentration
AUC0→inf | up to 72 hours post-administration
  Area under the plasma concentration-time curve from 0 h to infinity
λz | up to 72 hours post-administration
  λz-Terminal elimination rate constant
Residual area (%) | up to 72 hours post-administration
  The residual areas were determined in % by the following equation: {(AUC0→inf - AUC0→last) /AUC0→inf}* 100. The unit is %.
t1/2 | up to 72 hours post-administration
  t1/2 -The terminal half-life

CONTACTS AND LOCATIONS:
Overall Officials: Vlad Udovytskyi, Study Chair — Joint Stock Company "Farmak"
Locations (1):
- Arab Pharmaceutical Industry Consulting/Pharmaceutical Research Unit, Amman, Jordan

IPD SHARING:
Plan to Share IPD: No